CLINICAL TRIAL: NCT01586416
Title: Intervention to Increase Chemotherapy Tolerance in Elderly Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lara Traeger, Assistant in Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R03CA157200-01A1 (NIH); 1R03CA157200-01A1 (NIH)
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Colonic Neoplasms
Keywords: Colonic neoplasms; Older adults; Psychosocial Intervention; Chemotherapy adherence
MeSH Terms: conditions — Colonic Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Intervention (Experimental): Brief behavioral intervention on 2-3 sessions of tailored cognitive-behavioral therapy to support chemotherapy adherence and well-being of patients completing chemotherapy for colon cancer.
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Two or three one-hour sessions of an individual behavioral intervention led by a doctoral-level licensed psychologist during the first 12 weeks of chemotherapy. Intervention addresses modifiable behaviors for managing chemotherapy challenges.

SUMMARY:
The purpose of this study is to develop and pilot test a behavioral intervention for elderly adults in treatment for colon cancer, to enhance their skills for managing the challenges of completing chemotherapy regimens. The investigators will assess feasibility and acceptability of the intervention, and explore preliminary efficacy of the intervention for reducing psychological distress and improving rates of optimal chemotherapy adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Verbal fluency in English
* Diagnosis of colon cancer
* Scheduled to initiate chemotherapy treatment for colon cancer

Exclusion Criteria:

* Active, unstable, untreated serious mental illness interfering with ability to participate
* Cognitive impairment interfering with ability to participate
* Receiving radiotherapy concomitant with chemotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Participant satisfaction with intervention structure, timing and content | At approximately 12 weeks post-baseline
  Participants rate acceptability of structure, timing and content of intervention using Likert-type response scales, and are also invited to provide brief qualitative feedback on opinions about intervention.
Number of participants who withdraw from study after enrollment | At approximately 12 weeks post-baseline

SECONDARY OUTCOMES:
Change from baseline in the Hospital Anxiety and Depression Scale | At approximately 12 weeks post-baseline
Change from baseline in the Symptom Distress Scale | At approximately 12 weeks post-baseline
  The 13-item Symptom Distress Scale (SDS)measures physical and psychological symptom-related distress.
Proportion of each chemotherapy component administered during the treatment regimen relative to the total planned amount | At approximately 24 weeks post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States